CLINICAL TRIAL: NCT05042843
Title: Effect of 5,25% Sodium Hypochlorite Enamel Deproteinization on the Initial Shear Bond Strength and Glue Penetration in the Enamel of Orthodontic Brackets Bonded With a Self-etching Primer: An In Vitro Study on Human Bicuspids.
Brief Title: Effect of Deproteinization on the Shear Bond Strength and Glue Penetration in the Enamel of Orthodontic Brackets
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL21_0534
Record Dates: First submitted 2021-09-01; First posted 2021-09-13 (Actual); Last update posted 2021-09-13 (Actual); Status verified 2021-09

CONDITIONS: Orthodontic Appliance Complication
Keywords: glue penetration; orthodontic brackets; self-etching bracket

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — NC
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study was to evaluate the effects of enamel deproteinization on the initial shear bond strength (SBS) and on the bracket/adhesive failure mode of orthodontic brackets bonded with a self-etching primer (SEP) as a primary objective. As secondary objective a Raman microscopy study was performed to assess the resin penetration into the enamel according to the three bonding protocols.

ELIGIBILITY:
Inclusion criteria:

- All patient with orthodontic treatment involving bicupids extractions

Exclusion criteria:

- Patients with damaged teeth

Ages: 12 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All patient with orthodontic treatment involving bicupids extractions
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-01-30 (Actual)

PRIMARY OUTCOMES:
Number of resistance to tearing of orthodontic brackets stuck to extracted premolars | 1 day
  Number of resistance to tearing of orthodontic brackets stuck to extracted premolars

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane BARTHELEMI, PhD, Study Director — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC